CLINICAL TRIAL: NCT05777772
Title: Deprescribing to Reduce Injurious Falls Among Older Adults With Dementia
Acronym: STOP-FALLS-D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Elizabeth Phelan, Professor: School of Medicine, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00015806; 3U54AG063546 (NIH)
Record Dates: First submitted 2023-02-03; First posted 2023-03-21 (Actual); Results first posted 2024-05-07 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Educational Intervention (Experimental): Educational Intervention
  Interventions: Behavioral: STOP Falls D Educational Intervention

INTERVENTIONS:
Behavioral: STOP Falls D Educational Intervention — This is one-arm, health-system embedded pragmatic pilot trial

SUMMARY:
STOP-FALLS-D is an educational intervention to inform and activate patients, their care partner(s), and their primary care providers to work together to reduce use of central nervous system (CNS) active medications and prevent adverse outcomes (falls and injuries) associated with their use.

DETAILED DESCRIPTION:
The study design is a pragmatic, one-arm pilot trial to test the feasibility and acceptability of implementing a deprescribing intervention with older people with dementia and their care partners in primary care. The intervention consists of patient-facing educational brochures on CNS-active medications and decision support for the primary care provider. Ethnic/minority groups will be over-sampled to ensure a diverse study sample.

ELIGIBILITY:
Older Adult Sample

Inclusion Criteria:

* Diagnosed dementia (dementia diagnosis code or prescription for dementia medication)
* Receiving primary care at a Kaiser Permanente Washington integrated group practice outpatient clinic
* Prescribed at least one CNS-active medication on a chronic (3 months or more) basis

Exclusion Criteria:

* Skilled nursing facility resident
* Current cancer diagnosis
* On hospice or palliative care

Care Partner Sample

Inclusion Criteria:

* Aged 18 years or older
* Self-identify as a care partner for the older adult with dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2023-02-22 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Phelan, MD, Principal Investigator — University of Washington
Locations (1):
- Kaiser Permanente Health Research Institute, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Care Partners: Persons who help care for the older person with dementia
Period: Overall Study
Arm/Group | Educational Intervention | Care Partners
Started | 114 | 9
Completed | 114 | 9 (The number of care partners completed is fewer than the number planned due to care partners being an indirect target of the intervention.)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Educational Intervention Group: Educational Intervention
  STOP Falls D Educational Intervention: This is one-arm, health-system embedded pragmatic pilot trial
- Care Partners: Care partners of older people with dementia
- Total: Total of all reporting groups
Arm/Group | Educational Intervention Group | Care Partners | Total
Number analyzed (Participants) | 114 | 9 | 123
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 3 | 10
  >=65 years | 107 | 6 | 113
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Exact age was not collected for care partners. Age categories were collected.
  years
    number analyzed (Participants) | 114 | 0 | 114
    (all) | 79.9 (9.1) |  | 79.9 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 6 | 88
  Male | 32 | 3 | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 6 | 0 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 99 | 9 | 108
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 4 | 0 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 114 | 9 | 123

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dementia With Medically Treated Falls
Description: Number of older adult participants with dementia with a fall-related healthcare visit
Time Frame: Through study completion, up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Educational Intervention
Number analyzed (Participants) | 114
Participants | 24

2. Secondary Outcome: Number of Participants With Dementia With All-cause Emergency Department Visits or Hospitalizations
Description: Number of older adult participants with dementia with an emergency department visit or hospitalization for any reason
Time Frame: Through study completion, up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Educational Intervention
Number analyzed (Participants) | 114
Participants | 29

3. Secondary Outcome: Number of Participants With Dementia With Skilled Nursing Facility Placement
Description: Number of older adult participants with dementia admitted to a skilled nursing facility
Time Frame: Through study completion, up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Educational Intervention
Number analyzed (Participants) | 114
Participants | 5

ADVERSE EVENTS:
Time Frame: 6 months after initial mailing date
Description: Adverse events data were collected only for the older adults with dementia.
Arm/Group | Educational Intervention
All-Cause Mortality (participants affected / at risk) | 6/114
Serious Adverse Events (participants affected / at risk) | 0/114
Other Adverse Events (participants affected / at risk) | 0/114

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-17): https://cdn.clinicaltrials.gov/large-docs/72/NCT05777772/Prot_SAP_000.pdf